CLINICAL TRIAL: NCT01748630
Title: Pain, Fentanyl Consumption, and Delirium in Children After Scoliosis Surgery: Dexmedetomidine Versus Midazolam
Brief Title: Effects of Dexmedetomidine on the Postoperative Experience in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Dr Mustafasaid, Assist. Prof., Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOTM_Anaesthesia_MSA1
Record Dates: First submitted 2012-11-30; First posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Failed Moderate Sedation During Procedure
Keywords: scoliosis, sedation, children, fentanyl consumption, pain
MeSH Terms: conditions — Scoliosis; Pain | interventions — Dexmedetomidine; Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine, Midazolam (Active Comparator): dexmedetomidine (group DEX); starting dose, 0.4 μg•kg-1•h-1,with intermittent fentanyl
  Interventions: Drug: dexmedetomidine; Drug: fentanyl
- Midazolam (Active Comparator): midazolam (group MDZ); starting dose, 0.1 mg•kg-1•h-1
  Interventions: Drug: Midazolam; Drug: fentanyl

INTERVENTIONS:
Drug: dexmedetomidine
  Arms: Dexmedetomidine, Midazolam
Drug: Midazolam
  Arms: Midazolam
Drug: fentanyl

SUMMARY:
Background: The study aim was to compare the efficacy of dexmedetomidine versus midazolam for sedation during the early postoperative period in children who underwent scoliosis surgery.

Methods: We performed a prospective, randomized trial in an intensive care unit (ICU) in a tertiary care center. In this study, 42 patients (American Society of Anesthesiology physical status I and II) who underwent scoliosis surgery were divided into 2 groups according to sedation protocols: group DEX (n = 22) and group MDZ (n = 20). Children (12-18 years) requiring mechanical ventilation underwent a continuous infusion of either dexmedetomidine (group DEX; starting dose, 0.4 μg•kg-1•h-1) or midazolam (group MDZ; starting dose, 0.1 mg•kg-1•h-1) with intermittent fentanyl, as needed. The efficacy of sedation was assessed using the Richmond Agitation Sedation Scale (RASS). Quality of pain relief was measured using the Numeric Visual Analog Scale (NVAS). During the arousal assessment, delirium was determined in patients in the RASS range of -2 to +1 using the Confusion Assessment Method for the ICU (CAM-ICU). Fentanyl consumption, incidence of delirium, NVAS scores, and hemodynamics were recorded postoperatively at 2, 4, 6, and 24 h in the ICU.

ELIGIBILITY:
Inclusion Criteria:

admittance to the ICU and a requirement of mechanical ventilation with an endotracheal tube.

Exclusion Criteria:

Patients who had a history of allergies to midazolam and/or dexmedetomidine; delirium, developmental delay, or mental retardation, as reported by parents; an American Society of Anesthesiologists classification greater than III; any known previous reactions to anesthesia; or a history of asthma or an anticipated difficult airway and concomitant disease (neuromuscular scoliosis or neurodegenerative disease) were excluded from the study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
fentanyl consumption | 1 hour
fentanyl consumption | 2 hours
fentanyl consumption | 4 hours
fentanyl consumption | 6 hours
fentanyl consumption | 24 hours

SECONDARY OUTCOMES:
incidence of delirium | 1, 2, 4 ,6 and 24 hours

OTHER OUTCOMES:
heart rate | 1, 2, 4 ,6 and 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)